CLINICAL TRIAL: NCT00011479
Title: Single Dose Pharmacokinetic Study of Abacavir in HIV-Infected Children and Adolescents
Brief Title: Blood Levels of Abacavir After One Dose in HIV-Infected Children and Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: P1018; 11653 (Registry Identifier: DAIDS ES); ACTG P1018; PACTG P1018
Record Dates: First submitted 2001-02-22; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Administration, Oral; Drug Administration Schedule; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Pharmacokinetics; abacavir
MeSH Terms: conditions — HIV Infections | interventions — abacavir

INTERVENTIONS:
Drug: Abacavir sulfate

SUMMARY:
The purpose of this study is to measure blood levels of abacavir in children and adolescents over a period of time following a single dose so that a dosage for adolescents can be determined.

Little is known about how abacavir is cleared by the body in adolescents. It has been shown that young children require a higher abacavir dose based on weight than adults. Older children, or adolescents, may not require as high a dose. This study may provide information as to whether the children's dose or the adult dose is better for HIV-infected adolescents.

DETAILED DESCRIPTION:
Pharmacokinetic differences between children and adults have resulted in recommended doses of abacavir based on weight that are higher for children than for adults. There are insufficient data to determine whether the pediatric or adult dose is more appropriate for HIV-infected adolescent patients. This study measures pharmacokinetic data for abacavir in the adolescent population so that an appropriate dosage can be determined.

Patients are evenly enrolled into 2 groups based on Tanner Stage. Group I patients are Tanner Stage 1 or 2 (pre-pubertal). Group II patients are Tanner Stage 3, 4, or 5 (pubertal). Each patient receives a single oral dose of abacavir given as the commercially available oral solution. Pharmacokinetic blood samples are collected before dosing and at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4, 6, and 8 hours post dose for abacavir concentrations.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 9 to 18 years of age.
* Are HIV-positive.
* Have a CD4 cell count above 200 cells/microL.
* Have a viral load (level of HIV in the blood) under 100,000 copies/ml.
* Have not changed their anti-HIV drugs for the 4 weeks before study entry.
* Are able to swallow study medications.
* Both males and females, agree to use a barrier method of birth control for 3 days after taking the abacavir dose for this study. (This study has been changed. In the earlier version, no birth control was needed.)
* Can be followed at a participating Pediatric AIDS Clinical Trials Unit (PACTU) for the entire study.
* Provide written consent of a parent or guardian, if under 18 years of age.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have liver or kidney problems, as shown by screening tests.
* Have medical or surgical problems that affect movement or absorption in the stomach or gut.
* Have an opportunistic (AIDS-related) or serious bacterial infection requiring medicine at the time of enrollment.
* Have any diseases (other than HIV infection) or other findings that, in the investigator's opinion, might make it harmful for the patient to be on the study.
* Have a history of chronic alcohol use.
* Fall outside of a certain weight range for their age.
* Are pregnant or breast-feeding.
* Are receiving or have received abacavir.
* Are receiving nonnucleoside reverse transcriptase inhibitors, including efavirenz, delavirdine, or nevirapine; hydroxyurea; mycophenylate; rifampin, rifabutin, anticonvulsants, or other drugs that affect the liver; or chemotherapy for active cancer.
* Have received interferons, interleukins, HIV or other vaccines, or experimental therapy within 30 days before entering the study.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24
Dates: Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence D'Angelo, Study Chair; John Rodman, Study Chair
Locations (24):
- United States (24):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Children's Hospital of L.A. (Pediatric), Los Angeles, California
  - Univ of California, San Diego, San Diego, California
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Med College of Georgia, Augusta, Georgia
  - The Med Ctr Inc, Columbus, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Children's Hosp of Boston, Boston, Massachusetts
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Metropolitan Hosp Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Columbus Children's Hosp, Columbus, Ohio
  - Med Univ of South Carolina, Charleston, South Carolina
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas